CLINICAL TRIAL: NCT01300052
Title: A Multicenter, Randomized, Double-Blind, 12-Week Study Of The Safety And Efficacy Of AN2728 Versus AN2728 Vehicle In The Treatment Of Patients With Mild-To-Moderate Plaque-Type Psoriasis
Brief Title: AN2728 Topical Ointment to Treat Mild-to-Moderate Plaque-Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN2728-PSR-204; C3291017 (Other: Alias Study Number)
Record Dates: First submitted 2011-02-17; First posted 2011-02-21 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Psoriasis
Keywords: psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Ointments

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AN2728 ointment, 2% (Experimental): AN2728 ointment, 2%
  Interventions: Drug: AN2728 ointment, 2%
- Ointment Vehicle (Placebo Comparator): Ointment Vehicle
  Interventions: Drug: Ointment Vehicle

INTERVENTIONS:
Drug: AN2728 ointment, 2% — AN2728 ointment, 2%, applied twice daily for 12 weeks
  Arms: AN2728 ointment, 2%
Drug: Ointment Vehicle — Ointment Vehicle, applied twice daily for 12 weeks
  Arms: Ointment Vehicle

SUMMARY:
The purpose of this study is to determine whether AN2728 topical ointment is a safe and effective treatment for mild-to-moderate plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stable mild-to-moderate plaque-type psoriasis involving 2-35% of total body surface area (BSA) excluding face, scalp, and genitals
* Willingness and ability to apply study medication as directed, comply with study instructions, and commit to attending all study visits
* Women of childbearing potential must agree to use contraception for the entire study period

Exclusion Criteria:

* Any dermatological conditions that could interfere with clinical evaluations
* Concurrent or recent use of certain topical or systemic medications without a sufficient washout period
* Significant confounding conditions as assessed by study doctor
* Participated in any other trial of an investigational drug within 30 days or participation in a research study concurrent with this study
* Use of lithium- or hydroxychloroquine-containing products (e.g., Plaquenil)
* Use of a beta-blocking medication (e.g., propranolol) if the dose has not been stabilized for at least 3 months
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-01-26 (Actual); Primary Completion 2011-06-06 (Actual); Study Completion 2011-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (10):
  - The Savin Center, New Haven, Connecticut
  - Dermatology Specialists, PSC, Louisville, Kentucky
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Karl G. Heine, MD Dermatology, Henderson, Nevada
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Dermatology Consulting Services, High Point, North Carolina
  - Oregon Medical Research Center, Portland, Oregon
  - DermResearch, Inc, Austin, Texas
  - J&S Studies, Inc., College Station, Texas
  - The Center for Skin Research, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- AN2728 Ointment, 2%: AN2728 ointment, 2% was applied topically twice daily to all psoriasis plaques within each participant for 12 weeks (84 days). Plaques were identified at Baseline (Day 1) by the investigator
- AN2728 Ointment, Vehicle: AN2728 ointment vehicle was applied topically twice daily to all psoriasis plaques within each participant for 12 weeks (84 days). Plaques were identified at Baseline (Day 1) by the investigator.
Period: Overall Study
Arm/Group | AN2728 Ointment, 2% | AN2728 Ointment, Vehicle
Started | 46 | 22
Completed | 40 | 19
Not Completed | 6 | 3
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all randomized participants who received the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | AN2728 Ointment, 2% | AN2728 Ointment, Vehicle | Total
Number analyzed (Participants) | 46 | 22 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 20 | 61
  >=65 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 34 | 13 | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Success in Physician's Global Assessment (PGA) of Disease Severity at Day 84
Description: PGA assessed severity of overall disease activity in participants. It was performed using a 6-point scale graded from 0 - 5, in which 0 = clear (no plaque elevation above normal skin level), 1 = almost clear (essentially flat with possible trace elevation), 2 = mild (slight but definite elevation of plaque above normal skin level), 3 = moderate (moderate elevation with rounded or sloped edges to plaque), 4 = severe (marked elevation with hard, sharp edges to plaque), 5 = very severe (very marked elevation with very hard, sharp edges to plaque). The success in PGA of disease severity was defined as a PGA score of '0 = clear' or '1 = almost clear', with at least 2-grade improvement in PGA from Baseline to Day 84.
Time Frame: Day 84
Population: ITT population included all randomized participants who received the study medication. Missing data was imputed using last observation carried forward (LOCF) method.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AN2728 Ointment, 2% | AN2728 Ointment, Vehicle
Number analyzed (Participants) | 46 | 22
percentage of participants | 17.4 [6.4 to 28.3] | 13.6 [0.0 to 28.0]
Statistical Analysis 1: Comparison: AN2728 Ointment, 2% vs AN2728 Ointment, Vehicle; Difference in percentage was calculated as values of AN2728 Ointment, 2% group minus values of AN2728 Ointment, Vehicle group; Test type: Superiority or Other; Difference in Percentage = 3.8, 95% CI 2-sided [-14.3 to 21.8]

2. Secondary Outcome: Percentage of Participants Who Achieved Success in Physician's Global Assessment (PGA) of Disease Severity at Days 14, 28, 42, 56, and 70
Description: PGA assessed severity of overall disease activity in participants. It was performed using a 6-point scale graded from 0 - 5, in which 0 = clear (no plaque elevation above normal skin level), 1 = almost clear (essentially flat with possible trace elevation), 2 = mild (slight but definite elevation of plaque above normal skin level), 3 = moderate (moderate elevation with rounded or sloped edges to plaque), 4 = severe (marked elevation with hard, sharp edges to plaque), 5 = very severe (very marked elevation with very hard, sharp edges to plaque). The success in PGA of disease severity was defined as a PGA score of '0 = clear' or '1 = almost clear', with at least 2-grade improvement in PGA from Baseline to Day 14, 28, 42, 56 and 70.
Time Frame: Day 14, Day 28, Day 42, Day 56, Day 70
Population: ITT population included all randomized participants who received the study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AN2728 Ointment, 2% | AN2728 Ointment, Vehicle
Number analyzed (Participants) | 46 | 22
percentage of participants
  Day 14 | 2.2 [0.0 to 6.4] | 0 [NA to NA] — 95% Confidence Interval was not evaluable as there were no participants who achieved success in PGA at the specified time point
  Day 28 | 8.7 [0.6 to 16.8] | 4.5 [0.0 to 13.2]
  Day 42 | 26.1 [13.4 to 38.8] | 18.2 [2.1 to 34.3]
  Day 56 | 21.7 [9.8 to 33.7] | 13.6 [0.0 to 28.0]
  Day 70 | 17.4 [6.4 to 28.3] | 13.6 [0.0 to 28.0]

3. Secondary Outcome: Change From Baseline in Percentage of Body Surface Area (%BSA) Involved With Psoriasis at Day 84
Description: Percentage of the total body surface area (BSA) involved with psoriasis was measured. Change from Baseline (Day 1) in percentage of BSA at Day 84 was reported.
Time Frame: Baseline (Day 1), Day 84
Population: ITT population included all randomized participants who received the study medication. Missing data was imputed using LOCF method.
Measure: Mean (Standard Deviation); unit: percentage of body surface area
Arm/Group | AN2728 Ointment, 2% | AN2728 Ointment, Vehicle
Number analyzed (Participants) | 46 | 22
percentage of body surface area | -2.1 (3.20) | -1.4 (3.22)

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Day 84 that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAE and non-SAE.
Time Frame: Baseline (Day 1) up to Day 84
Population: Safety population included all randomized participants with confirmed usage of the study medication.
Measure: Number; unit: participants
Arm/Group | AN2728 Ointment, 2% | AN2728 Ointment, Vehicle
Number analyzed (Participants) | 46 | 22
participants
  AEs | 23 | 12
  SAEs | 0 | 2

5. Secondary Outcome: Number of Treatment-Emergent Adverse Events (TEAEs) by Severity
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs were classified according to the severity in 3 categories a) mild =AEs does not interfere with participant's usual function b) moderate =AEs interfered to some extent with participant's usual function c) severe =AEs interfered significantly with participant's usual function and required systemic drug therapy. Treatment-emergent were events between first dose of study drug and up to Day 84 that were absent before treatment or that worsened relative to pretreatment state. In this outcome measure, number of mild, moderate and severe TEAEs were reported.
Time Frame: Baseline (Day 1) up to Day 84
Population: Safety population included all randomized participants with confirmed usage of the study medication.
Measure: Number; unit: adverse events
Arm/Group | AN2728 Ointment, 2% | AN2728 Ointment, Vehicle
Number analyzed (Participants) | 46 | 22
adverse events
  Mild | 14 | 11
  Moderate | 25 | 5
  Severe | 5 | 5

6. Secondary Outcome: Number of Participants With Local Tolerability Symptoms: Burning/Stinging
Description: Local tolerability in participants was evaluated in terms of presence and absence of burning/stinging symptom and its severity in the areas of body where medication was applied. Burning/stinging symptoms were graded on a 4-point scale of 0 - 3 where 0 =none (no stinging/ burning), 1 =mild (slight warm, tingling sensation), 2 = moderate (definite warm; tingling/stinging sensation), 3 = severe (hot, tingling/stinging sensation that caused definite discomfort). Higher scores=Severe symptoms. In this outcome measure, number of participants with none, mild, moderate and severe burning/stinging symptoms were reported.
Time Frame: Baseline (Day 1) up to Day 84
Population: Safety population included all randomized participants with confirmed usage of the study medication. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | AN2728 Ointment, 2% | AN2728 Ointment, Vehicle
Number analyzed (Participants) | 40 | 19
participants
  None | 31 | 18
  Mild | 5 | 1
  Moderate | 4 | 0
  Severe | 0 | 0

7. Secondary Outcome: Number of Participants With Local Tolerability Symptoms: Pruritus
Description: Local tolerability was evaluated in participants in terms of presence and absence of pruritus symptom and its severity in the areas of body where medication was applied. Pruritus symptoms were graded on a 4-point scale of 0 - 3 where 0 =none (no pruritus), 1 =mild (occasional, slight itching/scratching), 2 = moderate (constant or intermittent itching/scratching which was not disturbing sleep), 3 = severe (bothersome itching/scratching which was disturbing sleep). Higher scores=Severe symptoms. In this outcome measure, number of participants with none, mild, moderate and severe pruritus symptoms were reported.
Time Frame: Baseline (Day 1) up to Day 84
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | AN2728 Ointment, 2% | AN2728 Ointment, Vehicle
Number analyzed (Participants) | 40 | 19
participants
  None | 23 | 13
  Mild | 8 | 6
  Moderate | 5 | 0
  Severe | 4 | 0

ADVERSE EVENTS:
Arm/Group | AN2728 Ointment, 2% | AN2728 Ointment, Vehicle
Serious Adverse Events (participants affected / at risk) | 0/46 | 2/22
Other Adverse Events (participants affected / at risk) | 23/46 | 12/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AN2728 Ointment, 2% (N=46) | AN2728 Ointment, Vehicle (N=22)
Cholecystitis infective (Infections and infestations) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AN2728 Ointment, 2% (N=46) | AN2728 Ointment, Vehicle (N=22)
Gastritis (Gastrointestinal disorders) | 1 | 0
Application site pain (General disorders) | 1 | 0
Application site pruritus (General disorders) | 1 | 0
Application site rash (General disorders) | 1 | 0
Medical device pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 1
Sinusitis (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 0
Guttate psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.